CLINICAL TRIAL: NCT02043925
Title: QT-prolongation in Psychiatric Hospitals
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Eline Vandael, PhD-student, KU Leuven
Other Study IDs: VF/2010/02
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: QT-prolongation
Keywords: QT-prolongation; Torsade de Pointes; drug interactions; psychiatry
MeSH Terms: conditions — Long QT Syndrome; Torsades de Pointes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- psychiatric patients treated with QT-prolonging drugs
  Interventions: Drug: drugs linked with QT-prolongation

INTERVENTIONS:
Drug: drugs linked with QT-prolongation — all the drugs that are mentioned in the lists of QT-prolonging drugs of CredibleMeds (www.crediblemeds.org)

SUMMARY:
Observational study in 6 psychiatric hospitals in Flanders. Patients are included when a QT-prolonging drug is added to a medication profile that already contains a potential QT-prolonging drug. An ECG is taken before the administration of the new drug and a week after starting the new drug to investigate the change in duration of the QTc-interval. Risk factors for developing QT-prolongation and blood concentrations of potassium and creatinine are documented.

ELIGIBILITY:
Inclusion Criteria:

* inpatient in one of the 6 participating psychiatric hospitals
* QT-prolonging drug in the medication profile and the doctor prescribes another QT-prolonging drug

Exclusion Criteria:

* age < 18 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational study in 6 psychiatric hospitals in Flanders. Patients are included when a QT-prolonging drug is added to a medication profile that already contains a potential QT-prolonging drug.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2010-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
change in QTc-interval (corrected for heart rate) | before and one week after the start of a QT-prolonging drug

CONTACTS AND LOCATIONS:
Overall Officials: Eline Vandael, PhD-student, Principal Investigator — KU Leuven
Locations (1):
- Psychiatrisch Centrum Sint-Jan, Eeklo, Belgium